CLINICAL TRIAL: NCT03074721
Title: PCI Suite: Road Map Fusion Imaging in Coronary Diagnostics and Therapy
Acronym: PCI Suite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-022
Record Dates: First submitted 2017-02-13; First posted 2017-03-09 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI with PCI Suite Software (Other)
  Interventions: Device: PCI Suite Software
- conventional PCI (Other)
  Interventions: Other: conventional PCI

INTERVENTIONS:
Device: PCI Suite Software — PCI with PCI Suite Software
  Arms: PCI with PCI Suite Software
Other: conventional PCI — conventional PCI without PCI Software
  Arms: conventional PCI

SUMMARY:
The PCI Suite is developed by Philips Medical Systems, a Philips Healthcare company. The proposed PCI Suite is a new software package which can be used during coronary interventions. The software package includes two sub-packages, known as StentBoost and Cardiac Roadmapping.

The patient will undergo standard of care medical treatment for his or her cardiac condition. During the procedure, the physician may make angiograms for diagnosis and as reference for device navigation as part of the standard care. These angiograms will be automatically processed in PCI Suite and displayed on fluoroscopy for navigation support. In case a balloon catheter is inserted into the coronary arteries, the physician may take cine images as part of the standard care. These images can be automatically enhanced in PCI Suite. The primary objective of this prospective, mono-center, randomized clinical trial is to evaluate the amount of contrast medium used during percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* hemodynamically relevant type A or B lesion

Exclusion Criteria:

* hemodynamically relevant type C lesion
* NSTEMI/STEMI
* declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Amount of contrast medium | Baseline
  Determination during PCI

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | Baseline, after 6 months, after 12 months
  Major adverse cardiac and cerebrovascular events (MACCE) are defined as occurence of myocardial ischemia, stroke, acute stent thrombosis, major bleeding
Procedural success | Baseline
  Defined by an open target vessel with a maximum of 20% residual stenosis and TIMI III flow
Procedure duration | Baseline
  Determination of duration of PCI
area dosage product | Baseline
  Determination during PCI

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Zeus, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quast C, Phinicarides R, Afzal S, Veulemans V, Klein K, Berisha N, Leuders P, Erkens R, Jung C, Bonner F, Kelm M, Polzin A, Zeus T. Roadmap fusion imaging in percutaneous coronary intervention reduces contrast medium exposure irrespective of investigator's experience level. J Invasive Cardiol. 2024 Jan;36(1). doi: 10.25270/jic/23.00203. PMID 38224296